CLINICAL TRIAL: NCT03540108
Title: The Cholesterol-lowering Efficacy of Probiotic Lactobacillus Plantarum ECGC 13110402 (LPLDL®) in Hypercholesterolemic Adults
Brief Title: The Efficacy of Cholesterol-lowering Probiotic Lactobacillus Plantarum LPLDL® in Hypercholesterolemic Adults.
Acronym: ProLoChol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Reader in Nutrition, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSC 18/ 241
Record Dates: First submitted 2018-04-30; First posted 2018-05-30 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; bile acid synthesis; cholesterol; bile salt hydrolysis; vitamin D; probiotic L plantarum LPLDL®
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, randomised, placebo-controlled, parallel-group design to determine the cholesterol-lowering efficacy of Lactobacillus plantarum ECGC 13110402 (LPLDL® in hypercholesterolaemic adults (>6mmol).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: L. plantarum ECGC 13110402 (LPLDL®) (Experimental): Lactobacillus plantarum ECGC 13110402 (LPLDL®) equivalent to 4 x10^9 CFU (0.1 g) with the addition of filling carrier (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed once a day, after lunch with 250mL of water.
  Interventions: Dietary Supplement: Lactobacillus plantarum ECGC 13110402
- Placebo Comparator: Maltodextrin (Placebo Comparator): Maltodextrin (an oligosaccharide without prebiotic effect) (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed once a day, after lunch with 250mL of water.
  Interventions: Dietary Supplement: Placebo Comparator: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum ECGC 13110402 — The study will consist of two phases: a treatment period (12 weeks) with either the active or placebo and a wash-out period (4 weeks). Following a screening visit to ensure adherence to the inclusion criteria, the study will consist of a baseline, midpoint, endpoint (week 6 and 12, respectively) and washout visit (week 16).
  Arms: Experimental: L. plantarum ECGC 13110402 (LPLDL®)
Dietary Supplement: Placebo Comparator: Maltodextrin — Please see intervention description above.
  Arms: Placebo Comparator: Maltodextrin

SUMMARY:
Coronary heart disease (CHD) is one of the major causes of death and disability in industrialised countries. Results from several epidemiological and clinical studies indicate a positive correlation between elevated total serum cholesterol levels, mainly reflecting the LDL-cholesterol fraction, and risk of CHD. It is thought that a reduction in total plasma cholesterol levels in populations suffering from primary hypercholesterolemia (elevated cholesterol) can lower the incidence of coronary thrombosis. Currently, therefore there is extensive interest in the management of serum cholesterol and other blood lipids. Diet is viewed as a major influencing factor that can reduce levels. This is largely driven by the expense of drug therapy, the large numbers of individuals affected and unwanted side effects of such treatments. Dietary strategies for prevention of CHD implicate adherence to a low-fat/low-saturated fat diet. Although such diets may present an effective approach, they are difficult to maintain on a long-term basis and efficacy diminishes over time. As such, new approaches towards identification of other dietary means of reducing blood cholesterol levels have been evaluated. These include, among others, the use of probiotics. Probiotics are 'live microbial feed supplements that offer a benefit to health'. They are marketed as health or functional foods whereby they are ingested for their purported positive advantages in the digestive tract and/or systemic areas like the liver, vagina or bloodstream. The main goal of the study is to test the efficacy of the probiotic in degrading cholesterol as well as produce metabolites that interfere with its synthesis in the liver in adults with high cholesterol (>6mmol). The effect may also be partially ascribed to an enzymatic deconjugation of bile acids.

DETAILED DESCRIPTION:
The aim of this human volunteer study is to establish the extent of extent of the cholesterol lowering potential of Lactobacillus plantarum ECGC 13110402 in 50 hypercholesterolaemic adults (35-70 years old).

ELIGIBILITY:
Inclusion Criteria:

* males and females from 35 to 70 years of age
* BMI 18.5 to 29.9 kg/m2
* total cholesterol (TC) >6mmol/L.

Exclusion Criteria:

* suffering from chronic gastrointestinal complaints (including chronic constipation, diarrhoea or Irritable Bowel Syndrome)
* diabetes or anaemia
* requirement to take long-term medications active on the gastrointestinal tract, treatment of cardio-vascular disease, or any other long-term medication
* high blood cholesterol or use of cholesterol lowering drugs/ functional foods
* history of drug or alcohol misuse or alcohol consumption exceeding 14 and 21 units/week for females and males respectively
* those suffering with any allergies to medication or food
* on weight-reducing diets.
* Females planning pregnancy within six months from the start of the study, lactating, or have given birth within the preceding six months
* use of antibiotics within six months preceding the study, participation in any probiotic, prebiotic or laxative study or intake of an experimental drug four weeks prior to the study start.
* Individuals exercising > 16 744 kJ per week

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Cholesterol-lowering efficacy | from baseline to 6 and 12 weeks of the intervention
  To test, in humans, whether the LPLDL® intervention lowers total cholesterol by a log change of min. 0.45 ± 0.4.
Effect on the gut microbiota | from baseline to 6 and 12 weeks of the intervention
  To determine the effect of LPLDL® on the faecal microbiota composition and microbial activity of the volunteers using DNA profiling from faeces (16s rRNA sequencing using Illumina MiSeq Platform and QIIME data analysis software).
Effect on vitamin D absorption and ABOB | from baseline to 6 and 12 weeks of the intervention
  To investigate the effect of LPLDL® on vitamin D absorption in the study population by measuring circulating vitamin D in blood using clinical chemistry and monitoring vitamin D intake from food diary.
Effect on bile acid metabolism | from baseline to 6 and 12 weeks of the intervention
  To assess any changes in bile acid metabolites and TMAO during the study trial using high performance liquid chromatography tandem mass spectrometry to analyse the urine samples.

SECONDARY OUTCOMES:
Digestive symptoms | from baseline to 6 and 12 weeks of the intervention
  Bristol diary form Bristol diary form.
Dietary assessment | from baseline to 6 and 12 weeks of the intervention
  To conduct an assessment of dietary intake in the study population using a validated four-day food diary and dietplan 7 dietary analysis software (Forestfield Ltd.)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Costabile, PhD, Study Director — University of Roehampton
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No